CLINICAL TRIAL: NCT06689358
Title: Thoracic Paravertebral Block for Postoperative Pain Management in PACU After VATS Surgeries: A Randomized Controlled Trial
Brief Title: Thoracic Paravertebral Block for Postoperative Pain Management After VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22 KHCC 158
Record Dates: First submitted 2024-11-06; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative
Keywords: Opioids, Pain Management,; Thoracic Paravertebral Block. VATS; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Arm 1: General anesthesia with TPVB; Type: Experimental Intervention: 0.4 ml/kg of 0.5% bupivacaine injected into the thoracic paravertebral space.
  Arm 2: General anesthesia alone (control group). Type: No intervention (control) Intervention: No intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia with TPVB (Experimental): 0.4 ml/kg of 0.5% bupivacaine injected into the thoracic paravertebral space
  Interventions: Drug: 0.4 ml/kg of 0.5% bupivacaine
- General anesthesia alone (control group). (No Intervention): General anesthesia SOC alone

INTERVENTIONS:
Drug: 0.4 ml/kg of 0.5% bupivacaine — 0.4 ml/kg of 0.5% bupivacaine injected into the thoracic paravertebral space
  Arms: General anesthesia with TPVB

SUMMARY:
This randomized controlled trial evaluated the efficacy of a thoracic paravertebral block (TPVB) in reducing opioid requirements and pain intensity in the PACU after video-assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
This randomized controlled trial evaluated the efficacy of a thoracic paravertebral block (TPVB) in reducing opioid requirements and pain intensity in the PACU after video-assisted thoracoscopic surgery (VATS). Adult patients scheduled for elective VATS who meet the eligibility criteria will be randomized to either Arm:

Arm 1: General anesthesia with TPVB;

Arm 2: General anesthesia alone (control group).

Primary Outcome: to assess Opioid requirement in the PACU

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective VATS, ASA physical status II-III, BMI 19-40.

Exclusion Criteria:

* Patient refusal, coagulation disorders, contraindications to TPVB, chronic analgesic use, mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Opioid requirement in the PACU | Opioid requirement assessed at 5 minutes, 15 minutes, 30 minutes post-PACU admission, and at PACU discharge (up to 4 hours)
  Opioid requirement in the PACU, recorded as "yes" or "no."

SECONDARY OUTCOMES:
Pain intensity measured by Numeric Rating Scale -NRS | Pain intensity measured using the Numeric Rating Scale (NRS) at 5 minutes, 15 minutes, 30 minutes post-PACU admission, and at PACU discharge (up to 4 hours)
  Pain intensity measured by Numeric Rating Scale- NRS at several time points, Range: 0 (no pain) to 10 (worst imaginable pain), Interpretation: Higher scores indicate worse pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Ahed Al-Edwan, MD, Principal Investigator — KHCC
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No